CLINICAL TRIAL: NCT06112639
Title: DANCE REhabilitation Experience (DANCEREX-DTx): Protocol for a Randomized Controlled Trial on Effectiveness of Digital Therapeutics in Chronic Neurological Disabilities
Brief Title: The DANCEREX Proof-of-Concept Study for Chronic Neurological Disorders
Acronym: DANCEREX-DTx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other); University of Milano Bicocca (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DANCEREX-DTx
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sclerosis, Multiple; Neurocognitive Impairment, Mild; Neurocognitive Dysfunction
Keywords: rehabilitation; multiple sclerosis; dementia; digital therapeutics; neurocognitive dysfunction; MRI; neuroinflammation; telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Lymphoma, Follicular; Cognition Disorders; Dementia; Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DANCEREX Treatment (Experimental): Multidimensional dance-based program with motivational support integrated into applied game. The treatment will last 12 weeks with a frequency of two sessions a week, each lasting about 45 min.
  Interventions: Device: DANCEREX-DTx
- Multidimensional dance-based program (Active Comparator): Multidimensional dance-based program without motivational support. The treatment will last 12 weeks with a frequency of two sessions a week, each lasting about 45 min.
  Interventions: Device: Multidimensional dance-based program
- Educational Program (Placebo Comparator): Educational/informative videos on managing of clinical conditions.The program will last 12 weeks with a frequency of two sessions a week, each lasting about 45 min.
  Interventions: Device: Educational Program

INTERVENTIONS:
Device: DANCEREX-DTx — DANCEREX treatment integrates the dance activities with an innovative motivational system into applied game
  The patients will perform the exercises (different dance styles, i.e., Irish Dance, Hip Hop, Cha Cha Cha) independently at home using videos that illustrate the activity to be performed for each treatment session on a mobile device (tablet). The intensity of the exercise will be moderate with a progressive increase in difficulty level over the weeks. The treatment will start with simple dance movements to be performed in a sitting position to proceed with gradually more complex sequences, always to be performed in safe conditions (first seated and then standing, holding onto a chair). In addition, the DANCEREX app involves a game dynamic in which the execution of the rehabilitation sessions "feeds" a digital book that allows the rehabilitation experience to be placed in a narrative context.
  Arms: DANCEREX Treatment
Device: Multidimensional dance-based program — Multidimensional dance-based program provided via a digital medicine telerehabilitation platform. The patient will perform the exercises (different dance styles, i.e., Irish Dance, Hip Hop, Cha Cha Cha) independently at home using videos that illustrate the activity to be performed for each treatment session on a mobile device (tablet). The intensity of the exercise will be moderate with a progressive increase in difficulty level over the weeks. The treatment will start with simple dance movements to be performed in a sitting position to proceed with gradually more complex sequences, always to be performed in safe conditions (first seated and then standing, holding onto a chair).
  Arms: Multidimensional dance-based program
Device: Educational Program — Subjects will view educational/informative videos on Tablet. The treatment will be provided via a digital medicine platform.
  Arms: Educational Program

SUMMARY:
The goal of this clinical trial is to test a new digital therapeutic solution which combines a holistic, multidimensional rehabilitation program based on dance and music with an innovative motivational system (DANCEREX-DTx) in Chronic Neurological Disorders (Multiple Sclerosis and pre-Mild Cognitive Impairment - MCI/ MCI at risk of Alzheimer's Disease). The main questions it aims to answer are 1] efficacy of the digital therapeutic solution in terms of adherence, clinical/functional measures, quality of life and surrogate measures; 2] usability and acceptability of the system.

Participants will be randomized (with an allocation ratio of 2:2:1) into the experimental group (DANCEREX - 24 sessions of multidimensional dance-based program integrated with an innovative motivational system), active comparator group (24 sessions of multidimensional dance-based program) and placebo group (24 sessions of educational program). Researchers will compare the experimental group to the other two groups to see if a digital therapeutic solution integrating a multidimensional dance-based program and motivational system is effective in increasing adherence to rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 85 years (adult and older adult);
2. education equal to or more than five years
3. agreement to participate with the signature of the informed consent form;
4. clinical diagnosis of Multiple Sclerosis (MS) according to the 2017 revised criteria of MC Donald - Expanded Disability Status Scale (EDSS) score equal or less than 4.5, R-R disease course, freedom from relapses, and steroid treatment for at least one month, OR clinical diagnosis of pre-Mild Cognitive Impairment - MCI (Subjective Memory Complaints and/or Subjective Cognitive Complaints)/MCI at risk of Alzheimer's Disease with the Clinical Dementia Rating (CDR) scale equal or less than 0.5
5. Normal score to a screening test for cognitive impairment (Montreal Cognitive Assessment test - MoCA test > 15.5 Santangelo et al., 2015)

Exclusion Criteria:

1. presence of comorbidities that prevent patients from undertaking a safe home program (e.g., balance problems, history of falls in the past 6 months, use of assistive devices for deambulation)
2. presence of overt hearing/visual impairment
3. for the MCI group, the absence of a caregiver/study partner able to support the participant;
4. no living in one's own home;
5. for the MS group, score in cerebellum function at EDSS greater than 3

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to treatment | 12 weeks of treatment
  Adherence to treatment, in terms of both numbers of drop-out and percentage of attended sessions on the total prescribed

SECONDARY OUTCOMES:
Change in global cognitive functioning and subdomains measured by Montreal Cognitive Assessment (MoCA; Conti et al., 2015) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  MoCA is a screening test for global cognitive functioning. It includes tasks involving several domains: visuospatial/executive function tests, naming, selective and sustained attention, language, abstraction, memory and orientation. High scores are indicative of better general cognitive performance.
Change in visuoperceptual and attentional abilities measured by Trail Making Test (TMT part-A and part-B; Giovagnoli et al., 1996) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  TMT is a neuropsychological test that involves visual scanning (TMT-A) and dual-task (TMT-B). The TMT is scored by how long it takes to complete each part of the test. High execution times indicate poor performance.
Change in visuoperceptual and attentional abilities measured by Symbol Digit Modalities Test (SDMT; Smith A., 1973; Nocentini U., 2006) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  This paper-pencil measure involves a substitution task using a coding key with nine different abstract symbols, each paired with a numeral. Below the key, a series of these symbols is presented, and the participant is asked to say the corresponding number for each symbol. The score consists of the number of correct substitutions within 90 seconds. Higher scores indicate better performance.
Change in executive functions, including visual attention and inhibitory control of behavior measured by Stroop Test (Caffarra et al., 2002) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The test consists of three consecutive parts that the subject must perform as quickly and accurately as possible: 1) read a list of color names on a sheet; 2) say the names of the colors of some colored spots on the sheet; 3) name the color of the ink with which the names of the colors were written. Two scores are calculated by summing the number of errors made and the time taken to complete all parts. High execution times and the number of errors indicate poor performance.
Change in Verbal and semantic fluency measured by The Verbal Fluency and Semantic Tests (Carlesimo et al., 1996; Novelli et al., 1986). | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The Verbal Fluency and Semantic Tests are neuropsychological tests to evaluate language skills and executive functions - lexical store size, lexicon access ability, and lexical organization. The verbal fluency test requires the participant to say all words starting with a certain letter in one minute. The test comprises three letters and the score is given by the number of correct words. The semantic fluency test requires participants to say all words of a semantic category in one minute. The test includes three semantic categories and the score is given by the amount of words. Higher scores are indicative of better performance.
Change in long term visual memory measured by Free and Cued Selective Reminding Test (FCSRT) (Frasson et al., 2011) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  FCSRT is a visual memory test that maximises encoding specificity. It assesses learning (immediate recall) and visual long-term (delayed recall) memory of visual stimuli. The administration is divided into three phases: 1) Encoding phase: naming of stimuli (three boards with four coloured stimuli each) and verification of encoding with cue; 2) Immediate recall phase: free immediate recall + recall with a cue for not recalled stimuli (this sequence is repeated three times with interference task between trials); 3) deferred recall phase (after 30 minutes of non-verbal tasks): free deferred recall + recall with a cue for not recalled stimuli. Six scores can be obtained: Immediate Free Recall (spontaneous recall in the three trials; range 0-36); Immediate Total Recall (total recall in the three trials - range 0-36); Delayed-Free Recall (range 0-12); Delayed Total Recall (range 0-12); Index of Sensitivity of Cueing (ISC) and Number of intrusions. Higher scores indicate better performance.
Change in long term verbal memory measured by 15-Words of Rey (Carlesimo et al., 1995) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  15-Words of Rey is a test for the assessment of learning and verbal long-term memory of new information. The test is divided into 3 parts: 1] 15 words are read to the subject. 2) immediate recall: at the end of the reading, the patient is asked to repeat as many words as possible in any order. This procedure is used with the same word list five consecutive times. 3) Delayed recall: after an interval of 15 minutes, during which visuospatial tests are performed, the patient is asked to remember as many words as possible from the list. Two scores can be obtained: Immediate Recall given by the sum of spontaneous recall in the the five trials (range 0-75) and Delayed Recall given by free deferred recall (range 0-15). Higher scores indicate better performance.
Change in Static and dynamic balance measured by Mini-Best Test (Franchignoni et al., 2010) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The Mini-BESTest aims to identify the disordered systems underlying the postural control responsible for poor functional balance. This tool is composed by 27 tasks (36 items in total) assessing bio-mechanical constraints, stability limits/verticality, anticipatory responses, postural responses, sensory orientation, and stability in gait. Each item is scored based on ordinal scale scoring from 0- 3 where 3 = best performances and 0 = worst performances. The total score is provided as a percentage. Higher scores are indicative of better performance.
Change in Aerobic Capacity and Gait measured by 6' Minute Walking Test (6MWT) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  6' Minute Walking Test (6MWT) is has been validated as a general indicator of overall physical performance and mobility for older people (Duncan et al 1993, Harad et al 1999). The total distance walked is measured.
Changes in affect measured by Positive-Negative Affect Schedule (PANAS; Watson et al, 1988) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The PANAS is a self-report questionnaire. The list is split up into two segments, or mood scales. One scale measures a person's positive emotion and the other scale measures the negative. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent agrees that this applies to him. The final score of the PANAS Scale / Positive and Negative Affect Schedule (PANAS) test is the sum of the 10 terms on the positive scale and the sum of the 10 terms on the negative scale. The value assigned is positive for answers on the positive scale and negative for answers on the negative scale.
Changes in Activation level of Patients measured by Patient Activation Measure 13 (PAM13; Hibbard et al., 2004) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  PAM13 is a 13-item scale that assesses a person's underlying knowledge, skills and confidence integral to managing his or her health and healthcare. PAM13 total score ranging from 0 to 100. Higher values represent a better outcome. Specifically, individuals in the lowest activation level do not yet understand the importance of their role in managing their health and have significant knowledge gaps and limited self-management skills. Individuals in the highest activation level are proactive with their health, have developed strong self- management skills, and are resilient in times of stress or change.
Changes in patient's self-rated health measured by EuroQol five dimensions (5D) and five levels (5L) (The EuroQol Group, 1990; Janssen et al.,2013) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  EQ-5D-5L is a measure of health status that consists of the EQ-5D descriptive system and of the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. A total of 3125 possible health states are defined, ranging from 1111 (no problems in all dimensions) to 5555 (extreme problems in all dimensions). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labeled 'The best health you can imagine' (scored as "100") and 'The worst health you can imagine' (scored as "0").
Changes in patient's self-rated health status measured by Short Form Health Survey 36 (SF36; Ware, 2000) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  SF-36 is a short scale on health status, consisting of 36 questions subdivided into eight scales: Physical Function, Physical Role, Body Pain, General Health, Vitality, Social Function, Emotional Role and Mental Health. Each scale is transformed into a 0-100 scale on the assumption that each question carries equal weight. A lower score indicates more disability.
Changes in patient's fatigue measured by Modified Fatigue Index Scale (MFIS; Kos et al., 2006) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  MFIS consists of 21 items on 5 points Likert scale (from 0 never to 4 always) to assess the physical, cognitive and psychosocial components of fatigue. Higher scores indicate a greater impact of fatigue on a person's activities.
Changes in depressive symptoms measured by Beck Depression Inventory for Primary Care (BDI-PC, Steer et al., 1999) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The BDI-PC is a 7-item questionnaire with each item rated on a 4-point scale (0-3). It is scored by summing ratings for each item (range 0-21). Higher scores indicate greater deflection of mood tone.
Changes in anxiety level measured by State-Trait Anxiety Inventory - Form Y (STAI - Y; Spielberger, 1983; Pedrabissi & Santinello, 1989) | Baseline, post-treatment (up to 12 weeks) and follow-up (up to 6 months from the baseline)
  The STAI-Y is a commonly used measure of trait and state anxiety (20 items for each). All items are rated on a 4-point scale (from "Almost Never" to "Almost Always"). STAI is scored by summing ratings for each item (State-Anxiety: range 0-80; Trait Anxiety: range 0-80). Higher scores indicate greater anxiety.

OTHER OUTCOMES:
Changes in brain morphometry as detected by Magnetic Resonance Imaging Examination. | Time Frame: Baseline, post-treatment (up to 12 weeks)
  T1weighted 3D images will be collected to test changes in brain morphometry
Changes in structural connectivity as detected by Magnetic Resonance Imaging Examination. | Time Frame: Baseline, post-treatment (up to 12 weeks)
  DWI sequences will be collected to detect changes in structural connectivity
Changes in functional connectivity as detected by Magnetic Resonance Imaging Examination. | Time Frame: Baseline, post-treatment (up to 12 weeks)
  Resting-State fMRI (Multi echo - Multi-Band) images will be collected for the assessment of brain activity at rest and functional connectivity.
Changes in inflammatory and anti-inflammatory cytokines as measured by blood sampling | Time Frame: Baseline, post-treatment (up to 12 weeks)
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the Inflammatory cytokines (TNF, IL1beta, TGF-beta, IL-6, IL-33, IL-8), and Anti-inflammatory cytokines (IL-10, IL-37),
Changes in protein associated to downstream inflammasome activation as measured by blood sampling | Time Frame: Baseline, post-treatment (up to 12 weeks)
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the protein associated to downstream inflammasome activation: IL-18, active-caspase-1(p20 kDa) for canonical NLRP3 activation and caspase- 4,5,8 for non-canonical NLRP3 activation.
Changes in neurotrophic and neuroendocrine factors as measured by blood sampling | Time Frame: Baseline, post-treatment (up to 12 weeks)
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the neurotrophic and neuroendocrine factors such as Brain-derived neurotrophic factor (BDNF), catecholamines (dopamine, noradrenaline, and adrenaline), serotonin, cortisol, acetylcholine and beta-endorphins
Changes in neurodegenerative marker as measured by blood sampling | Time Frame: Baseline, post-treatment (up to 12 weeks)
  The sera will be collected, centrifuged, stored, frozen at -80 C degrees, and shipped (when necessary) to the chosen sample-processing center. The serum will be used to measure by Enzyme-Linked ImmunoSorbent Assay (ELISA) and by Automated Immunoassay System (ELLA) the neurodegenerative marker such as Neurofilament-light chain (NFL)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pia Amato, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (3):
- Italy (3):
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - IRCCS Centro Neurolesi Bonino-Pulejo, Messina
  - IRCCS Fondazione Don Carlo Gnocchi ONLUS, Milan

REFERENCES:
- [Derived] Borgnis F, Blasi V, Realdon O, Mantovani F, Cotelli M, Manenti R, Campana E, Lo Buono V, Marino S, Mavrodiev PA, Saresella M, Trimarchi PD, Alberoni M, Amato MP, Baglio F. DANCE Rehabilitation EXperience (DANCEREX-DTx): Protocol for a randomized controlled trial on effectiveness of digital therapeutics in chronic neurological disabilities. Digit Health. 2025 Mar 25;11:20552076251324448. doi: 10.1177/20552076251324448. eCollection 2025 Jan-Dec. PMID 40144043
- See also: internet page of Institution — http://www.dongnocchi.it/ricerca-scientifica/i-centri-irccs/irccs-s-maria-nascente-milano/caditer
- See also: internet page of Research Unit — http://caditer.dongnocchi.it/